CLINICAL TRIAL: NCT05966454
Title: Complex And Simple Appendicitis: REstrictive or Liberal Post-operative Antibiotic eXposure (CASA RELAX) Using Desirability of Outcome Ranking (DOOR) and Response Adjusted for Duration of Antibiotic Risk (RADAR) -A Randomized Controlled Trial
Brief Title: Complex And Simple Appendicitis: REstrictive or Liberal Post-operative Antibiotic eXposure - UCSF
Acronym: CASA RELAX
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 21-35457
Record Dates: First submitted 2023-06-30; First posted 2023-07-28 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Appendicitis
MeSH Terms: conditions — Appendicitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Restricted Post-Operative Antibiotics Group (Experimental): Participants undergoing standard of care (SOC) with simple appendicitis will not receive post-operative antibiotics.
  Participants undergoing standard of care with complicated (gangrenous or perforated) appendicitis will receive up to 24 hours of SOC post-operative antibiotics.
  Interventions: Drug: Multiple standard of care antibiotics for appendicitis, at physicians' discretion
- Liberal Post-Operative Antibiotics Group (Active Comparator): Participants undergoing standard of care with simple appendicitis will receive 24 hours of post-operative SOC antibiotics
  Participants undergoing standard of care with complicated (gangrenous or perforated) appendicitis will receive 4 days of post-operative SOC antibiotics.
  Interventions: Drug: Multiple standard of care antibiotics for appendicitis, at physicians' discretion

INTERVENTIONS:
Drug: Multiple standard of care antibiotics for appendicitis, at physicians' discretion — Standard of Care Antibiotic use will be restricted to none or up to 24 hours of post-operative antibiotics.
  Arms: Restricted Post-Operative Antibiotics Group
Drug: Multiple standard of care antibiotics for appendicitis, at physicians' discretion — Standard of Care Antibiotic use will be permitted for 24 hours or up to 4 days of post-operative antibiotics.
  Arms: Liberal Post-Operative Antibiotics Group

SUMMARY:
The purpose of this study is to demonstrate the safety, efficacy, and feasibility of short-course post-operative antibiotic treatment for simple and complicated appendicitis

DETAILED DESCRIPTION:
This is a single center, randomized controlled trial to determine if decreasing the amount of antibiotics after appendicitis surgery can decrease the risk of adverse effects associated with antibiotics while at the same time ensuring participant safety.

ELIGIBILITY:
Inclusion Criteria:

Age ≥ 18 years

* Age ≥ 18 years
* Planned appendectomy (laparoscopic or open)
* Working telephone number or reliable method to contact patient after hospital discharge

Exclusion Criteria:

* Unable to consent
* Pregnant Women
* Prisoners
* Immunocompromised as determined by clinical team, or patients actively receiving steroids, chemotherapy, or immunosuppressing medications (for example tacrolimus), or patients with active hematologic malignancy affecting the immune system, leukopenia, or end-stage AIDS
* Heart failure
* Allergy to bupivacaine
* Unlikely to comply with treatment or follow-up
* Inpatient consultation for appendicitis
* Clinically suspected of sepsis based on Sepsis-3 definition
* Current use of antibiotics for other indications
* Type 1 Diabetes or uncontrolled hyperglycemia
* Surgeon preference
* Patient preference
* Research team unavailable

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Estimated)
Dates: Start 2023-06-06 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Infectious/Antibiotic Complications | Up to 30 days after appendicitis surgery
  Infectious/antibiotic complication requiring antibiotic treatment only, Emergency Department visit, hospital readmission, percutaneous drainage, and operative intervention as assessed by treating physician.
Number of participant deaths | Up to 30 days after appendicitis surgery
  Up to 30 days after appendicitis surgery

CONTACTS AND LOCATIONS:
Overall Officials: Lucy Kornblith, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- Zuckerberg San Francisco General Hospital, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Patient data will be shared with Denver health and combined with data from other independent sites for final analysis
Supporting Information: Study Protocol
Time Frame: Beginning 9 months and ending 36 months following article publication
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee identified for this purpose